CLINICAL TRIAL: NCT05082246
Title: Impact of Complimentary and Alternative Practices on Patient Wellbeing During Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Mihir Modi, Family Medicine Physician, WellSpan Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1659000
Record Dates: First submitted 2021-06-15; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Anxiety; Depression; Stress; Pain; Heart Rate; Blood Pressure
Keywords: Complementary; Alternative; Emotional Freedom Technique; Conscious Breathing; Heartfulness Meditation; Rehabilitation; Tapping; Meditation; Anxiety; Depression; Stress; Pain
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain

STUDY DESIGN:
Intervention Model Description: This study is a pilot designed to assess the quality of experience of patients measured through standardized assessment forms and objective parameters such as vital signs including blood pressure and heart rate. Participants will be compared with their own data for each intervention.
  This will be a prospective pilot pre-post study for the duration of eight weeks, or as long as required to obtain 30 participants. If, prior to the study, measurements of blood pressure and heart rate; pain scale ratings; and anxiety, depression and stress scale scores in patients show an overall improvement when compared to the same information taken after the completion of eight week weeks, then it can be concluded that these CAM methods are feasible and beneficial in the rehab setting.
Masking Description: No masking. All participants will be getting interventions and measurements will be taken pre- and post- intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre- and Post- Intervention (Other): Data will be gathered in participants with pre-intervention and post-intervention comparison.
  Interventions: Other: Conscious Breathing; Other: Heartfulness Meditation; Other: Emotional Freedom Technique

INTERVENTIONS:
Other: Conscious Breathing — During the Conscious Breathing session, participants will be asked to sit comfortably and with gently closed eyes. Participants will be guided through several different kinds of breathing techniques, where the will focus will be on the expansion of the chest or abdomen, releasing all tension from the body, and visualizing breathing light into the body.
Other: Heartfulness Meditation — During the Heartfulness Meditation session, participants will be asked to sit comfortably and with gently closed eyes. Starting with the feet and working towards the head, participants will be asked to relax each part of the body. Then participants will focus on the heart and imagine it filled with light and love. Participants will sit in this relaxed state for a few minutes to allow all stress and cares to be released.
Other: Emotional Freedom Technique — During the Emotional Freedom Technique session, participants will be asked to tap lightly on several acupressure points while saying a variety of statements regarding pain, anxiety, depression or stress. As participants tap on the acupressure points, participants will repeat phrases of affirmation and acceptance, and also talk through how pain, anxiety, depression or stress may cause distress but can learn to release these feelings. participants will be given a picture of where each of the acupressure points lie on the face, chest or head, and will also be given a script of what to say while tapping on each acupressure point. In addition, participants will be given a description of what each acupressure point "means" - its associated organ and what emotion that point helps to release.
  Other Names: EFT; Tapping

SUMMARY:
The study's objective is to assess whether CAM methods are feasible and beneficial in the WSRH setting; to assess stress (using the Perceived Stress Scale-14 and using BioSquares™), anxiety (using the Generalized Anxiety Disorder-7 scale), depression (using the Patient Health Questionnaire-9 scale), pain (using the Wong-Baker FACES scale), and vital signs using a multidisciplinary complementary approach with Heartfulness Meditation, Conscious Breathing, and Emotional Freedom Technique - the CAM practices for this study; and, to assess and compare the above scores for each participant just prior to and immediately after each treatment session.

The study hypothesizes that using CAM modalities in the WSRH is both feasible and beneficial in that patient population; the patients receiving the CAM modalities of treatment will show an improvement in the above-mentioned scores compared to participant scores prior to the intervention; and there may also be an improvement in patients' vital signs following the intervention of CAM practices.

DETAILED DESCRIPTION:
Acute inpatient rehabilitation programs mainly focus on improving the physical wellbeing of the patients with physical and occupational therapies. While these may also have an impact on the mental and emotional wellbeing of the patients, there is not much available as therapies for mental and emotional wellbeing in these patients. In this study, the investigators wish to assess the impact of a structured CAM model practice for patients in rehabilitation program. These services will be offered through trained professionals. Depression and anxiety, stress, sleep, vital signs such as heart rate, blood pressure and pain scores will be studied within the period of study.

The study's objective is to assess whether CAM methods are feasible and beneficial in the WSRH setting; to assess stress (using the Perceived Stress Scale-14 and using BioSquares™), anxiety (using the Generalized Anxiety Disorder-7 scale), depression (using the Patient Health Questionnaire-9 scale), pain (using the Wong-Baker FACES scale), and vital signs using a multidisciplinary complementary approach with Heartfulness Meditation, Conscious Breathing, and Emotional Freedom Technique - the CAM practices for this study; and, to assess and compare the above scores for each participant just prior to and immediately after each treatment session.

The study hypothesizes that using CAM modalities in the WSRH is both feasible and beneficial in that patient population; the patients receiving the CAM modalities of treatment will show an improvement in the above-mentioned scores compared to participant scores prior to the intervention; and there may also be an improvement in patients' vital signs following the intervention of CAM practices.

ELIGIBILITY:
Inclusion Criteria:

* Meets age requirement
* Willing to participate

Exclusion Criteria:

* Patients who are unwilling to participate in the study will be excluded.
* Patients who are unable to sit for 30 minutes due to either physical or mental conditions will be excluded.
* Patients with an active diagnosis or history of bipolar disorder, schizophrenia or post-traumatic stress disorder (PTSD), as determined by the WSRH physiatrists or psychologists will be excluded.
* Patients with active suicidal thoughts and who are being referred for mental health help will also be excluded.
* Patients with a Montreal Cognitive Assessment (MOCA) greater than 20 will be excluded.
* Patients will be excluded who have a history of schizophrenia, schizoaffective disorder, or other primary psychotic disorder, or dysthymia with onset before age 20; current substance use or abuse disorder, eating disorder, obsessive compulsive disorder (OCD), bipolar disorder, acute psychosis, schizophrenia or schizoaffective disorder, cognitive disorder, organic brain damage or mental disorder, pervasive developmental disorder, mental retardation, borderline personality disorder, persistent antisocial behavior, a primary diagnosis of a personality disorder or risk of suicide, chronic depression/dysthymia, major depressive episode, depression secondary to a concurrent medical disorder, and clinically relevant neurological/ somatic illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-25 (Estimated)

PRIMARY OUTCOMES:
Improvement in anxiety | Through completion of study, approximately 8 weeks
  Measurement of anxiety using the Generalized Anxiety Disorder-7 scale. The GAD-7 total score for the seven items ranges from 0 to 21, with 0 to 4 indicating minimal anxiety, 5 to 9 indicating mild anxiety, 10 to 14 indicating moderate anxiety, and 15 to 21 indicating severe anxiety
Improvement in depression | Through completion of study, approximately 8 weeks
  Measurement of depression using the Patient Health Questionnaire-9. PHQ-9 total score for the seven items ranges from 0 to 27, with 1 to 4 indicating minimal depression, 5 to 9 indicating mild depression, 10 to 14 indicating moderate depression, 15 to 19 indicating moderately severe depression, and 20 to 27 indicating severe depression.
Improvement in perceived stress | Through completion of study, approximately 8 weeks
  Measurement of perceived stress using Perceived Stress Scale 14 can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress; scores ranging from 14-26 would be considered moderate stress; and scores ranging from 27-40 would be considered high perceived stress.

SECONDARY OUTCOMES:
Improvement in heart rate | Day of intervention, approximately 6 hours
  Measurement of heart rate using pulse oximetry device.
Improvement in blood pressure | Day of intervention, approximately 6 hours
  Measurement of blood pressure using DynaMap device.
Improvement in skin temperature | Day of intervention, approximately 6 hours
  Measurement of skin temperature using BioSquares™. These adhesive squares are placed on the webbing of participants' skin between the thumb and forefinger. Skin temperature will change the color of the square. Black is temperature of 79 degrees Fahrenheit and indicates tenseness. Red is temperature of 74 degrees Fahrenheit and indicates nervousness. Green is temperature of 87 degrees Fahrenheit and indicates calmness. Blue is temperature of 791 degrees Fahrenheit and indicates a relaxed state.
Improvement in pain level | Day of intervention, approximately 6 hours
  Measurement of pain using Wong-Baker FACES scale. "No Hurt" is a pain score of zero. "Hurts Little Bit" is a pain score of two. "Hurts Little More" is a pain score of four. "Hurts Even More" is a pain score of six. "Hurts Whole Lot" is a pain score of eight. "Hurts Worst" is a pain score of ten. Each rating has a correlating facial expression.

CONTACTS AND LOCATIONS:
Overall Officials: Mihir Modi, DO, Principal Investigator — WellSpan Health
Locations (1):
- Wellspan Surgery and Rehabilitation Hospital, York, Pennsylvania, United States